CLINICAL TRIAL: NCT05011942
Title: Irrisept Spinal Fusion Pilot Study Protocol
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 146827
Record Dates: First submitted 2021-07-30; First posted 2021-08-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lumbar Spine Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomized 1:1 treatment of placebo or standard of care irrigation and Irrisept solution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- normal saline control arm (Placebo Comparator): ii. normal saline used after initial skin incision prior to coming through fascia, after placement of instrumentation (screws, hooks), prior to placement of bone graft, and after fascial closure iii. Irrigation exposure/soak time to be 1 min for each irrigation time point.
  Interventions: Device: Irrisept Irrigation solution
- Irrisept irrigation solution (Active Comparator): ii. Irrigation (Irrisept vs control of normal saline) used after initial skin inicision prior to coming through fascia, after placement of instrumentation (screws, hooks), prior to placement of bone graft, and after fascial closure iii. Irrigation exposure/soak time to be 1 min for each irrigation time point. iv. 1 bottle (450 mL) Irrisept irrigation to be used during case with normal saline rinse to follow at each irrigation time point in study subjects
  Interventions: Device: Irrisept Irrigation solution

INTERVENTIONS:
Device: Irrisept Irrigation solution — ii. Irrigation (Irrisept vs control of normal saline) used after initial skin inicision prior to coming through fascia, after placement of instrumentation (screws, hooks), prior to placement of bone graft, and after fascial closure iii. Irrigation exposure/soak time to be 1 min for each irrigation time point. iv. 1 bottle (450 mL) Irrisept irrigation to be used during case with normal saline rinse to follow at each irrigation time point in study subjects v. Normal saline irrigation will be used alone in control subjects at the same time points.

SUMMARY:
Study objectives include assessing the use of Irrisept irrigation solution in lumbar spinal fusion procedures and effect on clinical and patient reported outcome measures. This includes assessing postoperative SSI as well as fusion rates in addition to patient reported outcome measures.

DETAILED DESCRIPTION:
This is a randomized controlled pilot study with a study size of 50 patients. Results will be utilized to plan a larger scale study. Background literature supports the use of chlorhexidine gluconate as an irrigation solution to decrease SSI although this has not been conducted in this population of patients (lumbar spine fusion) to date. A decrease in SSI with Irrisept, could support the possible use of this as an irrigation solution to decrease infections postoperatively. It will be important to know the effect if any of Irrisept on fusion rates. This study will provide valuable information that may assist in future treatment and prevention of SSI in lumbar spinal fusion patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85, undergoing primary lumbar spinal fusion (less than or equal to 3 levels)

Exclusion Criteria:

* Prior lumbar fusion (decompression only okay), spinal infection, spinal neoplasm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative surgical site infections | assessed for change at 1 month
  Postop SSI
Postoperative surgical site infections | assessed for change at 3 months
  postop SSI
Postoperative surgical site infections | assessed for change at 6 months
  postop SSI
Postoperative surgical site infections | assessed for change at 12 months
  postop SSI

SECONDARY OUTCOMES:
Fusion rates after surgery | assessed at 1 month
  fusion rates after surgery with irrisept vs saline irrigation
Fusion rates after surgery | assessed for change at 3 months
  fusion rates after surgery with irrisept vs saline irrigation
Fusion rates after surgery | assessed for change at 6 months
  fusion rates after surgery with irrisept vs saline irrigation
Fusion rates after surgery | assessed for change at 12 months
  fusion rates after surgery with irrisept vs saline irrigation
Patient outcome measures | assessed at 1 month
  Visual Analog Score for pain measuring patient outcomes in both study arms
Patient outcome measures | assessed at 3 months
  Visual Analog Score for pain measuring patient outcomes in both study arms
Patient outcome measures | assessed at 6 months
  Visual Analog Score for pain measuring patient outcomes in both study arms
Patient outcome measures | assessed at 12 months
  Visual Analog Score for pain measuring patient outcomes in both study arms
Patient outcome measures | assessed at 1 month
  Oswestry Disability Index Questionnaire measuring patient outcomes in both study arms
Patient outcome measures | assessed at 3 months
  Oswestry Disability Index Questionnaire measuring patient outcomes in both study arms
Patient outcome measures | assessed at 6 months
  Oswestry Disability Index Questionnaire measuring patient outcomes in both study arms
Patient outcome measures | assessed at 12 months
  Oswestry Disability Index Questionnaire measuring patient outcomes in both study arms
Patient outcome measures | assessed at 1 month
  Scoliosis Research Society (SRS) 22 Questionnaire measuring patient outcomes in both study arms
Patient outcome measures | assessed at 3 months
  Scoliosis Research Society (SRS) 22 Questionnaire measuring patient outcomes in both study arms
Patient outcome measures | assessed at 6 months
  Scoliosis Research Society (SRS) 22 Questionnaire measuring patient outcomes in both study arms
Patient outcome measures | assessed at 12 months
  Scoliosis Research Society (SRS) 22 Questionnaire measuring patient outcomes in both study arms

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No